CLINICAL TRIAL: NCT06934187
Title: eFficacy Of Carpal tUnnel releaSe (FOCUS) - Protocol for Randomised Controlled Multicentre Triple-Blinded Placebo Surgery Carpal Tunnel Release Trial With Observational Group
Brief Title: Carpal Tunnel Release Efficacy Trial
Acronym: FOCUS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 89/2024
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Carpal Tunnel Syndrome (CTS); Carpal Tunnel Surgery
Keywords: Carpal tunnel syndrome; Carpal tunnel release; Placebo surgery; Sham surgery; Randomized controlled trial
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: This trial is a multicentre, multinational, randomised, controlled, triple-blinded superiority trial with 1:1 parallel groups. Participants in one group will undergo carpal tunnel release while those in the other group will undergo placebo surgery.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTR surgery (Active Comparator): Carpal tunnel release will be performed.
  Interventions: Procedure: Carpal tunnel release
- Placebo surgery (Placebo Comparator): Only skin incision will be performed.
  Interventions: Procedure: Placebo surgery

INTERVENTIONS:
Procedure: Carpal tunnel release — The operating surgeons will make a skin incision distally from the distal wrist crease and ulnar to the thenar crease. The appropriate tissues, including the subcutaneous tissue, palmar fascia, flexor retinaculum, and antebrachial fascia, will then be divided in CTR group. Haemostasis will be achieved using bipolar coagulation. The skin will be closed, and an appropriate dressing will be applied.
  Arms: CTR surgery
Procedure: Placebo surgery — Only an skin incision will be made and the same time as CTR operation takes will be waited until skin closure. An appropriate dressing will be applied.
  Arms: Placebo surgery

SUMMARY:
Background Carpal tunnel syndrome (CTS) is a prevalent condition that affects 2.7% of the population, especially women. It arises due to compression of the median nerve in the wrist and is linked to factors like diabetes, obesity, and physical workload. Non-surgical treatments such as splinting and corticosteroid injections are often the first approach for mild to moderate CTS but show mixed long-term results. Surgical intervention, carpal tunnel release (CTR), is frequently necessary and has a success rate of 75-88%. CTR is a safe procedure, but like any surgery, it carries risks, including scarring and nerve injury.

Rationale Despite its widespread use, the effectiveness of CTR surgery has not been rigorously tested through randomised controlled trials (RCT) against placebo. This leaves a critical gap in understanding whether observed improvements result from surgery or the natural course of CTS, which can sometimes resolve on its own. Previous RCT in hand surgery have faced methodological issues, emphasising the need for high-quality research to validate the benefits of CTR surgery.

Objectives

FOCUS (eFficacy Of Carpal tUnnel release) trial, aims to provide robust evidence of CTR's effectiveness compared to placebo. The null and alternative hypotheses of the trial are as follows:

* Null Hypothesis: The treatment effect of CTR is not superior to placebo surgery.
* Alternative Hypothesis: The treatment effect of CTR is superior to placebo surgery

Trial Design This multinational, triple-blinded RCT includes two groups: one receiving CTR and the other undergoing placebo surgery. An additional observational cohort will enhance the trial's generalisability. Recruitment begins in Finland, with plans to expand to Denmark, China and Australia. Experienced hand surgeons will perform all procedures, and the study adheres to rigorous international guidelines (SPIRIT).

Methods Eligible participants are screened and randomised 1:1 to receive either CTR or placebo surgery. In CTR, surgeons relieve pressure on the median nerve through a small incision. Placebo surgery involves a similar incision without addressing the nerve compression. Both procedures use the same pre- and post-operative care protocols to maintain participant blinding.

Data collection involves comprehensive patient assessments at six months, one, two, and five years. A validated tool, the 6-CTS scale, is the primary outcome measure, while secondary measures include nerve conduction tests, hand strength, and patient-reported satisfaction.

The study includes 96 participants, allowing for statistical analysis with 80% power to detect meaningful differences in outcomes.Trial is triple-blinded ensuring that participants, outcome assessors, and investigators remain unaware of treatment assignments, minimising bias. Patients will be randomly assigned to 1:1 parallel groups using an internet-based randomisation program.

Ethical considerations The trial complies with the Declaration of Helsinki and national regulations. Participants provide informed consent and can withdraw at any time.

Data Management and Safety Data is securely stored in compliance with GDPR, and interim analyses are conducted to monitor safety. An independent Data Safety and Monitoring Committee (DSMC) oversees the trial, reviewing any serious adverse events.

Expected Outcomes and Significance

Discussion The trial seeks to determine whether CTR surgery provides superior outcomes compared to placebo, addressing a critical gap in evidence for this common procedure. By including patient-reported outcomes and rigorous blinding, the study emphasises improvements that matter most to individuals with CTS.

This research has far-reaching implications for patients, surgeons, and policymakers, offering insights into the value of CTR surgery. The results could refine treatment guidelines, ensuring that surgical interventions are evidence-based and benefit those most in need.

Conclusion The FOCUS-trial represents a significant step forward in validating the effectiveness of CTR surgery. By setting a high standard for surgical research, it aims to provide clarity on a widely performed procedure, contributing to improved care and outcomes for individuals with CTS worldwide.

ELIGIBILITY:
Inclusion Criteria:

* CTS diagnosed with ENMG, Symptoms typical for CTS, Ability to understand and answer the questionnaires, ≥ 18 years old.

Exclusion Criteria:

* Recurrent CTS; Ongoing systematic steroid treatment, chemotherapy, or immunomodulatory treatment; Pregnancy or breast feeding; Intrinsic muscle atrophy; Peripheral neuropathies; and Profound cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
CTS-6 | Preoperative vs 1 year. Secondary time points 6 months, 2 years and 5 years
  The 6-item Carpal Tunnel Syndrome Symptoms Scale questionnaire (6-CTS) is a CTS-specific instrument addressing pain and numbness in daily living. 6-CTS gives a value between 1 (best) and 5 (worst).

SECONDARY OUTCOMES:
ENMG | Preoperatively and 1 year
  Electroneuromyography (ENMG) has been adopted as a standard procedure when diagnosing CTS, and it can help to track improvements in nerve conduction postoperatively.
EQ-5D-3L | Preoperatively, 6 months, 1 year, 2 years, 5 years
  EuroQoL 5-Dimension 3-Level (EQ-5D-3L) is a Quality-of-Life assessment tool, validated in multiple languages. Scores value usually between 1.00 (perfect health) and 0 (death), but a minimum value obtainable is -0.594 (health condition worse than death). Higher score is better.
VAS for pain | Preoperative, 6 months, 1 year, 2 years, 5 years
  Visual analogue scale (VAS) has been validated for pain evaluation. Values range from 0 to 100mm, higher is worse.
VAS for nocturnal numbness | Preoperative, 6 months, 1 year, 2 years, 5 years
  Visual analogue scale (VAS) has been used for evaluation of numbness after CTR. Values range from 0 to 100mm, higher is worse.
2-PD | Preoperatively, 6 months, 1 year
  Two-point discrimination (2-PD) has been shown to improve after CTR.
Grip, tripod grasp, and pinch strength | Preoperatively, 6 months, 1 year
  Grip, tripod, and pinch strength have been shown to increase after CTR
Willingness for a re-treatment | 1 year
  Willingness for a re-treatment will be assessed using the question: ""Would you prefer the same treatment again, if the result would be the same as it is now?" Possible answers are "Yes" and "No". Yes is a better answer and No is a worse answer.
Global rating | Preoperatively, 6 months, 1 year, 2 years, 5 years
  Patient-rated global improvement will be assessed using the question: "How would you rate the function and pain of your hand compared to the situation before the treatment?" Participants will provide responses on a 7-step Likert scale, ranging from "Much worse" to "Much better."
Adverse events | 6 months, 1 year, 2 years
  Adverse events will be recorded and monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Susanna B Hiltunen, MD, Principal Investigator — Wellbeing services county of North Savo, Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Northern Savonia, Finland

IPD SHARING:
Plan to Share IPD: Yes
Pseudonymised patient level data can be shared within the EU/ETA. Anonymous patient level data will be available globally. These include all gathered data. Data will be shared after the trial has been finished.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Protocol will be published during 2025. SAP will be published with the protocol. ICF will be uploaded to clinicaltrials.gov. Primary results will be published in a peer-reviewed journal in 2030. Analytic code will be submitted with the results.
Access Criteria: Data will be shared to researchers who provide a methodologically sound proposal. Proposals should be directed to mikko.raisanen@pshyvinvointialue.fi

DOCUMENTS (1):
  • Informed Consent Form (2025-01-05): https://cdn.clinicaltrials.gov/large-docs/87/NCT06934187/ICF_000.pdf